CLINICAL TRIAL: NCT02456116
Title: Efficiency Study About the Effect of Acupunctur on Postoperative Pain After Total Knee Arthroplastry
Brief Title: Efficiency Study About the Effect of Acupuncture on Postoperative Pain After Total Knee Arthroplasty
Acronym: APOPKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical Scientific Fund of the Mayor of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard M Hobusch, Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KP13067BGMPOA
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- acupuncture/PCA/NSAID (Experimental): standard program with defined points:
  1. Ear acupuncture needles bitten once (day 0-5)
  2. Body acupuncture, once a day 20 minutes (day -1/ 0/ 2/ 4), depth of the prick 0.5 - 1 cm, with DeQI feeling/sensation is released
  Interventions: Device: acupuncture/PCA/NSAID
- sham acupuncture/PCA/NSAID (Sham Comparator): standard program with defined points:
  1. Ear sham-acupuncture needles bitten once (day 0-5)
  2. Body sham-acupuncture, once a day 20 minutes (day -1/ 0/ 2/ 4), depth of the prick 0.5
  Interventions: Device: sham acupuncture/PCA/NSAID
- PCA/NSAID (Other): minimal intervention (included in every arm) standard boli of morphine by pressing a button of PCA availability in the postoperative period (day 0-4) readout once a day NSAID (non-steroid antiinflammatory drug) 2x i.v. (75mg diclofenac-sodium, 30 mg orphenadrine citrate) (day 0-4)
  Interventions: Other: PCA/NSAID

INTERVENTIONS:
Device: acupuncture/PCA/NSAID — standard program with defined points:
  1. Ear acupuncture needles bitten once (day 0-5)
  2. Body acupuncture, once a day 20 minutes (day -1/ 0/ 2/ 4), depth of the prick 0.5 - 1 cm, with DeQI feeling/sensation is released
  Arms: acupuncture/PCA/NSAID
Device: sham acupuncture/PCA/NSAID — standard program with defined points:
  1. Ear acupuncture needles bitten once (day 0-5)
  2. Body acupuncture, once a day 20 minutes (day -1/ 0/ 2/ 4), depth of the prick 0.5
  Arms: sham acupuncture/PCA/NSAID
Other: PCA/NSAID — standard boli of morphine by pressing a button of PCA
  Arms: PCA/NSAID

SUMMARY:
The purpose of this study is to evaluate the use of needle acupuncture in comparison to a conventional postoperative pain management in terms of reducing pain and pain medication use in an interdisciplinary setting in a controlled, randomized study design after implantation of total knee arthroplasty .

DETAILED DESCRIPTION:
1. Patients and Methods

   1.1 All patients will be treated at the Medical University of Vienna and receive a TKA due to advanced gonarthrosis. The study includes male and female patients. Every patient who is admitted for a TKA ( Total knee arthroplasty) implant is invited to take part in the study. Exclusion criteria: renal insufficiency, cardial insufficiency, coronary heart disease, use of morphines, hydrocodones, benzodiazepines before surgery.

   1.2 The acupuncture is carried out using sterile disposable acupuncture needles, steel with a copper coil, size 0.25 x 30 mm by experienced acupuncturists and students in their third training year of the post graduate TCM (traditionel chinese medicine) training course of the Medical University of Vienna. The standard acupuncture was compiled as a traditional Chinese conventional body and ear/auricular acupuncture by a consortium of acupuncture professors as follows: Body acupuncture, pricked from both sides, the depth of the prick 0.5 - 1 cm, according to the technique of traditional Chinese acupuncture a DeQI (a sensation in the area of the acupuncture or in the course of the corresponding meridian) released. Regarding the frequency: ear acupuncture needles are bitten only postoperatively and can be left for a period of 4 until 7 postoperative days . The body acupuncture needling is carried out at the points of question once a day for a period of about 20 minutes , starting at the first preoperative day, continuating the day of surgery and 2nd and 4th postoperative day.

   In sham acupuncture the given acupuncture points are pricked 2-3 centimetres from the defined point.

   The group of patients who is not receiving any acupuncture and only used the PCA (Patient Controlled Analgesia) pain pump therapy is chosen as a control group. The pain pump therapy is not the subject of this clinical study and is routinely used for postoperative pain in TKA operations and does not need any evaluation.

   1.3 Randomising

   Patients who agree to take part in the study are randomised and blinded for the surgeon into 3 groups regarding the planned pain therapy.

   For postoperative pain therapy all patients receive, an on demand pain pump with morphine with controlled amounts of analgesics. The groups were formed on the assumption of a 30% reduction of pain using acupuncture in a power analysis with α=…… assuming 3 groups with 30 people each.: The method of randomising occurs as a sequence.

   The blinding applied especially to the surgeon and the patients who received real and sham acupuncture.
2. Outcome measures:

The primary aim is to find out if additive pain therapy in the form of body and ear/auricular acupuncture can effectively prove pain reduction after TKA implantation.

The amount of applied analgesics on every postoperative day (1.-5.) defines the command variable. The efficiency of acupuncture should be measured accordingly to the reduction of the on demand pain pump therapy.

Secondary objectives are the VAS of every postoperative day (1.-5.), the assessment of the operated leg's mobility as well as peri-operative nausea.

The intensity of pain is recorded as follows:

A) indirectly using the protocol of the amount of morphine administered by the PCA pump B) measuring pain by VAS (routinely 3 x daily)

ELIGIBILITY:
Inclusion Criteria:

* patients with advanced osteoarthritis of the knee (primary and secondary reasons)
* planned surgical procedure TKA

Exclusion Criteria:

* renal insufficiency
* cardial insufficiency
* coronary heart disease
* regular therapeutic use of morphines, hydrocodones, benzodiazepines before surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Amount of morphines/day | 1.-4.day postoperative
  Morphine PCRA (pain pump) administered to every patient

SECONDARY OUTCOMES:
movement abilities | 1.-4.day postoperative
  range of motion/Knee society score
Quality of Life (QOL) | day -1/day 5
  SF36 (short form 36)
Pain intensity (VAS) | 1.-4.day postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard M Hobusch, Dr., Principal Investigator — Medical University of Vienna, Department of Orthopaedics
Locations (1):
- Vienna General Hospital, Vienna, Austria

REFERENCES:
- [Background] Lin JG, Chen WL. Review: acupuncture analgesia in clinical trials. Am J Chin Med. 2009;37(1):1-18. doi: 10.1142/S0192415X09006679. PMID 19222107
- [Background] Wang JF, Bao HX, Cai YH, Zhang JH, Tong PJ. [Case-control study on application of auricular acupuncture for the treatment of analgesia during perioperative period in total hip arthroplasty]. Zhongguo Gu Shang. 2012 Mar;25(3):220-3. Chinese. PMID 22712373
- [Background] Usichenko TI, Kuchling S, Witstruck T, Pavlovic D, Zach M, Hofer A, Merk H, Lehmann C, Wendt M. Auricular acupuncture for pain relief after ambulatory knee surgery: a randomized trial. CMAJ. 2007 Jan 16;176(2):179-83. doi: 10.1503/cmaj.060875. PMID 17224599